CLINICAL TRIAL: NCT02609074
Title: Pilot Clinical Trial of CPC/rhBMP-2 Microffolds as Bone Substitute for Bone Regeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East China University of Science and Technology (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai 6th People's Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Yuan Yuan, Professor, East China University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFDA No.(2013):3460199
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Bone Fracture
Keywords: bone substitute; CPC; rhBMP-2
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPC/rhBMP-2 (Experimental): All operations were done by doctors titled with associate chief physician or above. Procedures were performed under general anesthesia in a tertiary care medical center.
  A minimally invasive internal fixation method had been applied in the surgeries. In brief, the patients with fracture were treated by reduction of fracture first of all, the correction of displacement, and the angle of the deformity, and the use of metal implants were fixed, and the collapse of the cancellous bone was filled with CPC/rhBMP-2 microffolds (product of Shanghai Rebone Biomaterials Co., Ltd, following the manufacturer's instruction), which was compacted and prevented from filling material into the joint cavity.
  Interventions: Procedure: Minimally invasive internal fixation surgeries; Device: CPC/rhBMP-2 micro-scaffolds
- CPC (Active Comparator): All operations were done by doctors titled with associate chief physician or above. Procedures were performed under general anesthesia in a tertiary care medical center.
  A minimally invasive internal fixation method had been applied in the surgeries. In brief, the patients with fracture were treated by reduction of fracture first of all, the correction of displacement, and the angle of the deformity, and the use of metal implants were fixed, and the collapse of the cancellous bone was filled with CPC paste (product of Shanghai Rebone Biomaterials Co., Ltd, following the manufacturer's instruction), which was compacted and prevented from filling material into the joint cavity.
  Interventions: Procedure: Minimally invasive internal fixation surgeries; Device: CPC paste

INTERVENTIONS:
Procedure: Minimally invasive internal fixation surgeries
Device: CPC/rhBMP-2 micro-scaffolds
  Arms: CPC/rhBMP-2
Device: CPC paste
  Arms: CPC

SUMMARY:
Objective: The investigators initiated a pilot clinical study to test safety and preliminary efficacy in humans (bone tissue repairing capacity) and to evaluate standard clinical and rehabilitation protocols.

Summary Background Data: Bone tissue engineering scaffolds loading growth factors have been considered as the most perspective among all bone substitutes, yet little progress of its clinical translation has been made. The concept of "micro-scaffolds" was proposed in this study to provide a trajectory to its clinical translation.

Methods: Pre-cured CPC/rhBMP-2 micro-scaffolds have been successfully developed and further applied as an easy-to-operate filler for bone regeneration in a pilot clinical study. Patients of tibial plateau fractures, proximal humeral fractures, or calcaneal fractures at a similar level of severity were randomly divided into two groups and treated by CPC/rhBMP-2 microffolds or traditional CPC paste (control group).

DETAILED DESCRIPTION:
Objective: The investigators initiated a pilot clinical study to test safety and preliminary efficacy in humans (bone tissue repairing capacity) and to evaluate standard clinical and rehabilitation protocols.

Summary Background Data: Bone tissue engineering scaffolds loading growth factors have been considered as the most perspective among all bone substitutes, yet little progress of its clinical translation has been made. The concept of "micro-scaffolds" was proposed in this study to provide a trajectory to its clinical translation.

Methods: Pre-cured CPC/rhBMP-2 micro-scaffolds have been successfully developed and further applied as an easy-to-operate filler for bone regeneration in a pilot clinical study. Patients of tibial plateau fractures, proximal humeral fractures, or calcaneal fractures at a similar level of severity were randomly divided into two groups and treated by CPC/rhBMP-2 microffolds or traditional CPC paste (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Age 16~70 years.
2. Tibial plateau fractures, proximal humeral fractures, or calcaneal fractures at a similar level of severity.
3. An understanding of the rehabilitation protocol and willing to follow it.
4. An agreement to postoperative visits and tests.
5. Signed an informed subject consent form.

Exclusion Criteria:

-

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
X-ray | Pre-operation; 1, 2, 3, 4, 6, 8, 12, 18 and 24 months post-operation.
  X-ray radiography at different time intervals after implantation was employed to observe the osseointegration of the implanted microffolds to host bone and the degradation of the material.
Clinical examination | 1 week post-operation
  The assessment was based on clinical examination. After the CPC implantation, all patients were observed according to the following indexes: allergic or toxic reactions, rash or high fever.

SECONDARY OUTCOMES:
Function scoring - IOWA knee score | 1, 2, 3, 4, 6, 8 and 12 months post-operation.
  The functional recovery was recorded at each follow-up time point using IOWA knee score in cases of tibial plateau fractures. The IOWA knee score is a questionnaire and clinical-examination-based evaluation of the function of the knee. The knee score is a five- category measurement, which includes activities of daily living, freedom from pain, gait, aid dependence, deformity and range of movement. The scores are grouped into excellent (90 to 100), good (80 to 89), fair (70 to 79) and poor (under 70) categories.
Function scoring - IOWA ankle score | 1, 2, 3, 4, 6, 8 and 12 months post-operation.
  The functional recovery was recorded at each follow-up time point using IOWA ankle score in cases of calcaneal fractures. The IOWA ankle score is a questionnaire and clinical-examination-based evaluation of the function of the ankle. The ankle score is a four-category measurement of function, freedom from pain, gait and range of movement. The scores are grouped into excellent (90 to 100), good (80 to 89), fair (70 to 79) and poor (under 70) categories.
Function scoring - NEER shoulder score | 1, 2, 3, 4, 6, 8 and 12 months post-operation.
  The functional recovery was recorded at each follow-up time point using Neer shoulder score in cases of proximal humeral fractures. Neer shoulder score has three parts: scoring of pain during the previous week by patients (verbal rating scale); clinical testing of function (muscle strength, reaching ability, and stability) and active range of motion; and an anatomical or radiological evaluation. The scores are grouped into excellent (90 to 100), good (80 to 89), fair (70 to 79) and poor (under 70) categories.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Liu, Ph.D., Study Chair — Engineering Research Center for Biomaterials of Ministry of Education, East China University of Science and Technology; Yuan Yuan, Ph.D., Principal Investigator — Engineering Research Center for Biomaterials of Ministry of Education, East China University of Science and Technology; Jinwu Wang, Ph.D., Principal Investigator — Ninth People's Hospital of Shanghai Jiao Tong University